CLINICAL TRIAL: NCT06439940
Title: Pilot Test for an Early Diagnosis Kit for Breast Cancer Based on Liquid Biopsies
Brief Title: Oncoliq: Early Breast Cancer Detection Based on Liquid Biopsies and microRNAs
Status: Recruiting | Type: Observational
Sponsor: Oncoliq US Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 459 EMnP0S0 / 21
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Female; Breast Cancer; Breast Carcinoma
Keywords: early diagnosis; early detection; cancer; breast cancer; miRNAs; liquid biopsies; pilot study; pilot test; liquid biopsy; Oncoliq; machine learning; AI; RT-qPCR
MeSH Terms: conditions — Breast Neoplasms; Disease; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women aged 50 to 70 who attend the gynecological annual check-up
  Interventions: Diagnostic Test: Blood sample extraction

INTERVENTIONS:
Diagnostic Test: Blood sample extraction — We do not alter the patient's regular gynecological check-up in any way. The patient will undergo a mammogram and a blood draw. We will then separate a small aliquot of blood for the purposes of the research protocol.

SUMMARY:
Oncoliq is a novel early breast cancer detection test based on liquid biopsies and microRNAs. This innovative test aims to improve the accuracy of cancer detection, thereby reducing patient mortality and healthcare costs.

To develop this test, the discovery and validation phases have been completed. In addition, Machine learning and AI were used to determine the algorithm for breast cancer detection.

The overall objective of this protocol is to implement a pilot test to enroll 1,000 women without a previous cancer diagnosis who are attending their annual medical check-up.

To achieve this, we will develop the following specific objectives:

Enroll women over age 35 who attend the gynecological annual check-up. Test the plasma of the enrolled volunteers for specific miRNA biomarkers using RT-qPCR.

Perform an analysis based on artificial intelligence techniques in collaboration with IMAGO Systems (USA) on mammogram images.

Compare the results obtained from the clinical check-up (BiRad from mammogram), IMAGO Systems and RT-qPCR (Oncoliq breast test). Conduct a 5-year follow-up on volunteers with pathological results from Oncoliq breast test.

Participants who meet the inclusion and exclusion criteria and agree to take part in the protocol will be required to sign both pages of the Informed Consent Form and complete the Annex and Survey. Subsequently, a small blood sample of 3-5 mL will be drawn via venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 35 years old who visit the gynecological clinic for their annual mammographic check-up

Exclusion Criteria:

* Personal history of cancer

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This protocol includes female volunteers over 35 years old with no personal history of oncological disease who visit the gynecology unit at "Hospital Posadas" for a gynecological and mammographic check-up.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
BIRADS mammography | From July 14 2021 to December 31 2024

SECONDARY OUTCOMES:
Level of miRNAs in blood sample detected with RT-qPCR | From March 2023 to December 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nacional Profesor Alejandro Posadas, El Palomar, Morón, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://meetings.asco.org/abstracts-presentations/237379